CLINICAL TRIAL: NCT01930318
Title: Effect of COX-2 Selective Inhibitors on Postoperative Insulin Resistance, Tramadol PCA and Early Postoperative Enteral Nutrition in Patients After Gastrointestinal Laparoscopic Surgery
Brief Title: Effect of COX-2 Selective Inhibitors on Postoperative Insulin Resistance After Gastrointestinal Laparoscopic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kong Wencheng, Senior Resident, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PTP-IR-EEN-1
Record Dates: First submitted 2013-08-25; First posted 2013-08-28 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PCA,Placebo,Placebo (Placebo Comparator): PCA for 2 days after operation, i.v placebo in 2 days after surgery and oral placebo in the day 3 to day 5 after surgery
- PCA,placebo,tramadol (Placebo Comparator): PCA for 2 days after operation, i.v placebo in 2 days after surgery, and oral tramadol in the day 3 to day 5 after surgery
- PCA,parecoxib,placebo (Experimental): PCA for 2 days after operation, i.v parecoxib in 2 days after surgery,and oral placebo in the day 3 to day 5 after surgery
  Interventions: Drug: parecoxib
- PCA,parecoxib,celecoxib (Experimental): PCA for 2 days after operation,i.v parecoxib in 2 days after surgery and oral celecoxib in the day 3 to day 5 after surgery
  Interventions: Drug: parecoxib

INTERVENTIONS:
Drug: parecoxib — 4 groups: PCA,Placebo,Placebo-PCA for 2 days after operation, i.v placebo in 2 days after surgery and oral placebo in the day 3 to day 5 after surgery; PCA,placebo,tramadol-PCA for 2 days after operation, i.v placebo in 2 days after surgery, and oral tramadol(0.1g t.i.d.) in the day 3 to day 5 after surgery;PCA,parecoxib,placebo-PCA for 2 days after operation, i.v parecoxib(40mg b.i.d.) in 2 days after surgery,and oral placebo in the day 3 to day 5 after surgery;PCA,parecoxib,celecoxib-PCA for 2 days after operation,i.v parecoxib(40mg b.i.d.) in 2 days after surgery and oral celecoxib(0.2g b.i.d.) in the day 3 to day 5 after surgery
  Other Names: COX-2 selective inhibitors
  Arms: PCA,parecoxib,celecoxib; PCA,parecoxib,placebo

SUMMARY:
It is well established that the resistance to the effects of insulin on glucose metabolism develops with a lot of stress hormone release after surgical trauma. This condition is known as insulin resistance (IR) characterized by hyperglycemia, hyperinsulinemia and lactic acidosis. Surgical IR not only affect glucose metabolism but also influence protein synthesis, then further exacerbate the depletion of the carbohydrate, fat and protein.

Postoperative pain is a challenging task for patients and surgeons, and it is part of the stress response to trauma and surgery, while the fear of pain can exacerbate the stress response.

The main aim of this study was to invest whether effective postoperative analgesia can reduce the stress response and insulin resistance.

ELIGIBILITY:
Inclusion criteria:

* Patients with gastrointestinal cancer scheduled for gastrointestinal laparoscopic surgery
* Patients between the ages of 18 and 70 yr
* ASA physical status I-II
* Requirements of informed consent and assent of participant, parent or legal guardian as applicable
* Consciousness and ability to cooperate

Exclusion criteria：

* History of alcohol, analgesic, or narcotic abuse
* Used analgesics, neuroleptics, antipsychotic agents, or corticosteroids within 6 hours of surgery
* A clinically significant laboratory abnormality or a history of significant cardiac, pulmonary, hepatic, or renal disease
* Female with positive pregnancy
* Allergy to conventional NSAIDs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance in perioperative period of gastrointestinal laparoscopic surgery | 5 days after operation

SECONDARY OUTCOMES:
The consumption of total and incremental tramadol after surgery. | 5 days after operation
The tolerated dose of enteral nutrition every day after surgery | 5 days after operation
Postoperative inflammatory factors (IL-4, IL-6 and TNF-α) and levels of stress hormone (glucocorticoids and catecholamines) in perioperative period of gastrointestinal laparoscopic surgery | 5 days after operation
Rest energy metabolism was measured in perioperative period to evaluate the caloric and substrate needs of our patients | 5 days after operation
The time of the first bowel movements and anal exhaust time after surgery | 5 days after operation or more
Pain intensity at rest and during leg raising recorded daily after surgery using Visible Numeric Rating Scale | 5 days after operation
Incidence of adverse events throughout the treatment period including nausea, vomiting, headache, urinary retention, somnolence, flatulence, and pruritus | 5 days after operation or more
Liver and renal function tests in perioperative period | 5 days after operation
Self-rating anxiety scale and self-rating questionnaire for depression before surgery | 1 day before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Kong, MD, Principal Investigator — Nanjing University
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Xu Z, Li Y, Wang J, Li J. Effect of postoperative analgesia on energy metabolism and role of cyclooxygenase-2 inhibitors for postoperative pain management after abdominal surgery in adults. Clin J Pain. 2013 Jul;29(7):570-6. doi: 10.1097/AJP.0b013e318270f97b. PMID 23328338